CLINICAL TRIAL: NCT06111521
Title: A PHASE 1 STUDY TO EVALUATE THE EFFECTS OF MULTIPLE DOSES OF LY3537982 ON THE SINGLE-DOSE PHARMACOKINETICS OF MIDAZOLAM, DIGOXIN, AND ROSUVASTATIN IN HEALTHY ADULT SUBJECTS
Brief Title: A Drug-Drug Interaction Study of LY3537982 on Midazolam, Digoxin, and Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-RAS-23007; J3M-OX-JZQJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3537982 + Digoxin & Rosuvastatin (Part 1) (Experimental): Single oral doses of digoxin and rosuvastatin with or without multiple doses of LY3537982 administered orally
  Interventions: Drug: LY3537982; Drug: Digoxin; Drug: Rosuvastatin
- LY3537982 + Midazolam (Part 2) (Experimental): Single doses of midazolam administered either orally or intravenously (IV) with or without multiple doses of LY3537982 administered orally
  Interventions: Drug: LY3537982; Drug: Midazolam

INTERVENTIONS:
Drug: LY3537982 — Administered orally
  Other Names: Olomorasib
Drug: Digoxin — Administered orally
  Arms: LY3537982 + Digoxin & Rosuvastatin (Part 1)
Drug: Rosuvastatin — Administered orally
  Arms: LY3537982 + Digoxin & Rosuvastatin (Part 1)
Drug: Midazolam — Administered orally
  Arms: LY3537982 + Midazolam (Part 2)
Drug: Midazolam — Administered IV
  Arms: LY3537982 + Midazolam (Part 2)

SUMMARY:
The main purpose of this study is to evaluate the effects of multiple doses of LY3537982 on the pharmacokinetics (PK) of digoxin (a P-glycoprotein [P-gp] substrate), rosuvastatin (a breast cancer resistance protein [BCRP)] substrate), and midazolam (a substrate of Cytochrome P450 3A4 [CYP3A4]) in adult healthy participants. The study will also evaluate the safety and tolerability of LY3537982 with or without single doses of digoxin, rosuvastatin, and midazolam. The study is conducted in two parts. Participants will stay in the research center during the study, which will last about 23 and 11 days for part 1 and part 2, respectively, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease
* Body mass index (BMI): 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Females who are lactating or of childbearing potential
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Part 1: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3537982 | Predose on day 11 up to day 17
  Part 1: PK: Cmax of LY3537982
Part 1: PK: Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC[0-inf]) of LY3537982 | Predose on day 11 up to day 17
  Part 1: PK: AUC[0-inf] of LY3537982
Part 1: PK: AUC from Time 0 to time of the last measurable concentration (AUClast) of LY3537982 | Predose on day 11 up to day 17
  Part 1: PK: AUClast of LY3537982
Part 1: PK: Cmax of Digoxin | Predose on day 1 up to day 21
  Part 1: PK: Cmax of Digoxin
Part 1: PK: AUC[0-inf] of Digoxin | Predose on day 1 up to day 21
  Part 1: PK: AUC[0-inf] of Digoxin
Part 1: PK: AUClast of Digoxin | Predose on day 1 up to day 21
  Part 1: PK: AUClast of Digoxin
Part 1: PK: Cmax of Rosuvastatin | Predose on day 1 up to day 21
  Part 1: PK: Cmax of Rosuvastatin
Part 1: PK: AUC[0-inf] of Rosuvastatin | Predose on day 1 up to day 21
  Part 1: PK: AUC[0-inf] of Rosuvastatin
Part 1: PK: AUClast of Rosuvastatin | Predose on day 1 up to day 21
  Part 1: PK: AUClast of Rosuvastatin
Part 2: PK: Cmax of LY3537982 | Predose on day 4 up to day 11
  Part 2: PK: Cmax of LY3537982
Part 2: PK: AUC[0-inf] of LY3537982 | Predose on day 4 up to day 11
  Part 2: PK: AUC[0-inf] of LY3537982
Part 2: PK: AUClast of LY3537982 | Predose on day 4 up to day 11
  Part 2: PK: AUClast of LY3537982
Part 2: PK: Cmax of Midazolam | Predose on day 1 up to day 9
  Part 2: PK: Cmax of Midazolam
Part 2: PK: AUC[0-inf] of Midazolam | Predose on day 1 up to day 9
  Part 2: PK: AUC[0-inf] of Midazolam
Part 2: PK: AUClast of Midazolam | Predose on day 1 up to day 9
  Part 2: PK: AUClast of Midazolam
Part 2: PK: Cmax of 1'-Hydroxymidazolam | Predose on day 1 up to day 9
  Part 2: PK: Cmax of 1'-Hydroxymidazolam
Part 2: PK: AUC[0-inf] of 1'-Hydroxymidazolam | Predose on day 1 up to day 9
  Part 2: PK: AUC[0-inf] of 1'-Hydroxymidazolam
Part 2: PK: AUClast of 1'-Hydroxymidazolam | Predose on day 1 up to day 9
  Part 2: PK: AUClast of 1'-Hydroxymidazolam

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, Study Director — Loxo Oncology, Inc.
Locations (1):
- ICON Early Clinical & Bioanalytical Solutions, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No